CLINICAL TRIAL: NCT00714116
Title: An Ascending Single Dose Study Of The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Sbi-087 Administered To Subjects With Systemic Lupus Erythematosus.
Brief Title: Study Evaluating The SBI-087 In Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Emergent Product Development Seattle LLC (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3227K2-1002; B2261004 (Other: Alias Study Number)
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: safety; pharmacokinetics
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — SBI-087

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBI-087 (Experimental)
  Interventions: Drug: SBI-087

INTERVENTIONS:
Drug: SBI-087 — Single IV or SC dose of SBI-087

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of SBI-087 in subjects with Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE (by greater than or equal to 4 American College of Rheumatology [ACR] Revised Criteria) greater than 6 months before study day 1.
* History of a positive antinuclear antibody (ANA) titer greater than or equal to 1:160 or equivalent.

Exclusion Criteria:

* Treatment with more than 20 mg of prednisone per day.
* Evidence of unstable clinically significant disease (e.g., cardiovascular, cerebrovascular, respiratory, or renal disease, or any other unstable serious disorder) other than SLE.
* History of cancer (other than resected cutaneous basal and squamous cell carcinoma or in situ cervical cancer) with less than 5 years' documentation of a disease-free state.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety (physical examinations, laboratory tests, adverse events) and tolerability (dose-limiting toxicities) of ascending single doses of SBI-087 in subjects with Systemic Lupus Erythematosus (SLE) | 12 months

SECONDARY OUTCOMES:
Initial pharmacokinetic and pharmacodynamic profiles of SBI-087 in subjects with Systemic Lupus Erythematosus (SLE) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Arthritis & Rheumatology Care Center, South Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - MRA Clinical Research, South Miami, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas

REFERENCES:
- [Derived] Cohen S, Clowse M, Pardo P, Bhattacharya I, Menon S, Gourley I, Diehl A. Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of SBI-087, a CD20-Directed B-cell Depleting Agent: Phase 1 Dose Escalating Studies in Patients With Either Mild Rheumatoid Arthritis or Systemic Lupus. Clin Ther. 2016 Jun;38(6):1417-1434.e2. doi: 10.1016/j.clinthera.2016.03.028. Epub 2016 Apr 21. PMID 27112532
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3227K2-1002&StudyName=Study%20Evaluating%20The%20SBI-087%20In%20Subjects%20with%20Systemic%20Lupus%20Erythematosus